CLINICAL TRIAL: NCT06634823
Title: Prospective Placebo-Controlled Trial of Intramuscular Steroid Administration for the Treatment of Unexplained Chronic Cough
Brief Title: Efficacy of Intramuscular Steroid Injection for Chronic Cough.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Lauren Howser, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00140403
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Cough (CC); Laryngeal Disease; Coughing
Keywords: Throat; Chronic cough; Neurogenic cough; Unexplained cough
MeSH Terms: conditions — Chronic Cough; Laryngeal Diseases; Cough | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo injection into deltoid (arm)
  Interventions: Drug: Saline injection
- Steroid (Experimental): Triamcinolone injection into deltoid (arm)
  Interventions: Drug: Triamcinolone Acetonide Injectable Suspension

INTERVENTIONS:
Drug: Triamcinolone Acetonide Injectable Suspension — Triamcinolone injection into deltoid muscle (arm)
  Arms: Steroid
Drug: Saline injection — Saline injection into deltoid muscle (arm)
  Arms: Placebo

SUMMARY:
The primary goal of this study is to test the hypothesis that injecting steroid intramuscularly is an effective treatment for unexplained chronic cough. This will be achieved through the design of a prospective, placebo-controlled, single-blind, randomized clinical trial in which one group of patients will undergo a steroid injection into the deltoid muscle and the second group will undergo a placebo injection into the deltoid muscle. Data to determine if a clinically significant difference exists between the outcomes of the two groups will be measured by a dichotomous yes/no response to improvement, the Leicester Cough Questionnaire, and a visual analogue scale for symptom severity. This will provide the answer to the general question of whether or not the intramuscular injections are clinically effective for patients with unexplained chronic cough. Furthermore, any adverse reactions will be thoroughly documented. If this hypothesized treatment is proven effective, this can greatly improve the care of chronic cough patients by allowing for an evidence-based treatment option and a treatment option that may improve access to care. While the superior laryngeal nerve (SLN) injection is typically performed by fellowship trained laryngologists, intramuscular injections could be more widely utilized by general otolaryngologists or providers in other fields of medicine.

DETAILED DESCRIPTION:
A significant subset of patients are found to have "unexplained chronic cough", which is a diagnosis of exclusion. For these patients, the etiology of the cough is often not isolated. However, the cause is thought to be related to hypersensitivity and inflammation of both the nerves involved in cough sensation and/or mucosa of the larynx. A similar theory described by Driessen et al. hypothesizes that neuroinflammation related to glial cells in central and peripheral neural pathways may contribute to chronic cough in a similar way to how chronic pain is mediated by this pathway. Glial cells in the central and peripheral nervous system may be an important target for steroid hormones and their metabolites, which may have impact on inflammation and excitatory action.

Superior laryngeal nerve injections have been well studied in literature and were recently studied here at the Medical University of South Carolina in a prospective placebo-controlled trial for use in neurogenic cough. This study showed that there was a significant improvement in cough compared to placebo. This study was completed using randomization of 17 patients into the control and steroid/lidocaine injection groups. In the treatment group, 80% of patients reported improvement in symptoms, while in the control group only 14% of patients reported improvement. The Leicester Cough Questionnaire (LCQ) and visual analog scoring were used to compare cough data from pre and post injection.

The hypothesis revolves around the idea that SLN blocks may actually work systemically, so the site of injection may not be the key in cough improvement. This combined with the theory on glial cell involvement and systemic steroid use to inhibit the neuroinflammatory pathway leads us to believe that intramuscular steroid injections could improve chronic cough. Therefore, this study focuses on the use of systemic intramuscular steroids in patients with chronic cough and we hypothesize that patients will have improvement in cough severity. By opening another treatment option that could be utilized by general (non-fellowship trained) otolaryngologists, access to care and treatment may be improved for patients with chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* History consistent with chronic unexplained or refractory cough
* Age ≥ 18

Exclusion Criteria:

* Current smokers
* Uncontrolled diabetes (A1c>7%)
* Patients on ACE inhibitors or Angiotensin II receptor blockers (ARBs)
* Abnormal pulmonary function testing (PFTs) since start of the cough
* Patients with uncontrolled obstructive sleep apnea
* Abnormal chest X-ray within past 6 months
* Uncontrolled reflux
* Prior superior laryngeal nerve injection
* Current neuromodulating medication use for chronic cough*

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Leicester Cough Questionnaire | 4 weeks
  The primary outcome for which this study is powered is the change in mean Leicester Cough Questionnaire (LCQ) scores, both global and specific domains (physical, psychological, and social) from baseline to 1-4 weeks post-treatment. This score will be 19-133, with higher score indicating better outcomes.

SECONDARY OUTCOMES:
Visual Analog Scale | 4 weeks
  Visual analog scale for symptom severity. This will be reported as a percentage (ratio of X marked spot to total line).
Dichotomous yes/no to symptom improvement | 4 weeks
  Yes/No response to cough improvement

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Howser, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD can be made available at the end of the trial with de-identified patient data. A data dictionary will be provided so that the data can be fully interpreted.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After trial completion for 1 year
Access Criteria: Qualified researchers from academic institutions will be able to request access by contacting the PI.